CLINICAL TRIAL: NCT06418607
Title: Phase 1, Open Label, Randomized, Single-center, 2-sequence, 2-period, 2 Treatment Single Dose Crossover Bioequivalence Study Comparing Venglustat Tablet Formulation (Test) to Hard Capsule Formulation (Reference)
Brief Title: A Study of the Safety, Tolerability, and Bioequivalence of Orally Administered Venglustat in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BEQ15920; U1111-1239-0220 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — venglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Venglustat hard capsule administered in period 1 followed by tablet administered in period 2.
  Interventions: Drug: Venglustat
- Sequence 2 (Experimental): Venglustat tablet administered in period 1 followed by hard capsule administered in period 2.
  Interventions: Drug: Venglustat

INTERVENTIONS:
Drug: Venglustat — Pharmaceutical form:Tablet-Route of administration:Oral
  Other Names: GZ/SAR402671
Drug: Venglustat — Pharmaceutical form:Hard Capsule-Route of administration:Oral
  Other Names: GZ/SAR402671

SUMMARY:
The purpose of this study is to assess the bioequivalent effect of venglustat in tablet and hard capsule form when give with water under fasting conditions. Also, to evaluate the safety and tolerability of a single dose tablet and hard capsule of venglustat (swallowed whole) under fasting conditions in healthy adult participants. The maximum duration for participants from screening is up to 47 days.

DETAILED DESCRIPTION:
Total study duration for participants is up to 47 days including screening up to 20 days, 1 day of treatment in period 1 of 8-10 days, 1 day of treatment in period 2 of 8 days and followed by a final observation over 7 days (+/- 2 days).

ELIGIBILITY:
Inclusion Criteria: -Body mass index between 18.0 and 30.0 kg/m2, inclusive.

* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Vital signs after 10 minutes resting in supine position within the following ranges:
* 95 mmHg < systolic blood pressure (SBP) <140 mmHg,
* 50 mmHg < diastolic blood pressure (DBP) <90 mmHg,
* 45 bpm < heart rate (HR) <100 bpm.
* Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position in the following ranges; 120 ms < PR <220 ms, QRS <120 ms, QTc ≤450 ms (Fridericia algorithm recommended), 45bpm < HR <100 bpm and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
* Laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for healthy participant. Serum creatinine, hepatic transaminases (aspartate aminotransferase, alanine aminotransferase), and alkaline phosphatase should not exceed 1.25X the upper laboratory norm. Total biluribin out of normal range can be acceptable if total bilirubin does not exceed 1.5 the upper limit with normal conjugated bilirubin values (unless the participant has documented Gilbert syndrome).
* Having given written informed consent prior to undertaking any study-related procedure.
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
* Not under any administrative or legal supervision or under institutionalization due to regulatory or juridical order.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Required to either practice true abstinence consistent with their preferred and usual lifestyle, or use double contraceptive methods for the entire duration of the treatment until 6 weeks after the last treatment with venglustat for women and until 90 days for men Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* Blood donation, any volume, within 2 months before inclusion.
* Presence or history of clinically significant drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis). Note that 12 fluid ounces of regular beer, 5 fluid ounces of wine, and 1.5 fluid ounces of distilled spirits each contain approximately 14 g of alcohol.
* Smoking regularly more than approximately 5 cigarettes or equivalent per week, unable to stop smoking during the study (occasional smoker can be enrolled). Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).
* If female, pregnancy (defined as positive β-HCG test) or breast-feeding.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion. Any drug which could impact by any mechanism of action, the pharmacokinetics of the investigational medicinal product, including moderate and strong CYP3A4 inhibitors or inducers.
* Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any participant enrolled or having participated, in any other clinical study involving an investigational medicinal product or in any other type of medical research, and is still in the exclusion period according to applicable regulations.
* Any participant who cannot be contacted in case of emergency.
* Any participant who is the Investigator or any subinvestigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study, or any person dependent (employees or immediate family members) on the study site, the investigator or the sponsor.
* Prisoners or participant who are legally institutionalized.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV-1 and anti HIV-2 Ab).
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Positive alcohol test.
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 5 days before inclusion).
* Any participant who cannot comply with the following study restrictions: refraining from drinking alcohol, tea, coffee, chocolate, quinine, or caffeine-containing beverages from 1 day before institutionalization and throughout the study duration; not smoking or using tobacco from 1 day prior to institutionalization throughout the study duration until the end of-study visit; following a stable lifestyle with no intensive physical activity from 1 day prior to institutionalization throughout the study duration until the end-of-study visit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration observed (Cmax) of venglustat | Multiple time points up to day 16
Area under the plasma concentration versus time curve calculated from time zero to the real time (tlast) (AUClast) of venglustat | Multiple time points up to day 16
Area under the plasma concentration versus time curve (AUC) of venglustat | Multiple time points up to day 16

SECONDARY OUTCOMES:
Number of participants with adverse events | Multiple time points up to day 47
Time to reach Cmax (tmax) of venglustat | Multiple time points up to day 16
Interval between administration time and the sampling time preceding the first concentration above the limit of quantification (tlag) of venglustat | Multiple time points up to day 16
Terminal half-life associated with the terminal slope (λz) (t1/2z) of venglustat | Multiple time points up to day 16
Apparent total body clearance of a drug from the plasma (CL/F) of venglustat | Multiple time points up to day 16
Apparent volume of distribution at steady state (Vss/F) of venglustat | Multiple time points up to day 16

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami Site Number : 8400001, Miami, Florida
  - Prism Research Site Number : 8400002, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org